CLINICAL TRIAL: NCT04623593
Title: Economic Evaluation of Anterior Cervical Discectomy With Arthroplasty Versus Anterior Cervical Discectomy With Fusion in the Surgical Treatment of Cervical Degenerative Disc Disease, a Randomized Controlled Trial
Brief Title: Cervical Arthroplasty Cost Effectiveness Study (CACES)
Acronym: CACES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valérie Schuermans (Other)
Responsible Party: Sponsor-Investigator, Valérie Schuermans, Coordinating Investigator, Zuyderland Medisch Centrum
Organization: Zuyderland Medisch Centrum (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL72534.096.20
Record Dates: First submitted 2020-09-29; First posted 2020-11-10 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Radiculopathy, Cervical; Myelopathy Cervical; Myelopathy, Compressive; Radiculopathy, Cervical Region; Radiculopathy; in Spondylosis; Radiculopathy; in Intervertebral Disc Disorder; Myelopathy Neurological; Myelopathy Due to Spondylosis; Cervical Disc Disease; Cervical Disc Herniation; Cervical Disc Degeneration; Cervical Disc Disorder With Myelopathy; Cervical Disc Prolapse With Myelopathy; Cervical Spondylosis; Cervical Fusion; Cervical Disc Disorder With Radiculopathy; Cervical Disc Prolapse With Radiculopathy; Fusion of Spine; Disc Prolapse Cervical
Keywords: Cost-effectivity; Economic evaluation; Health Utility; Randomised controlled trial; RCT; ACDA; ACDF; Anterior cervical discectomy and fusion; Anterior cervical discectomy with arthroplasty; Degenerative cervical myelopathy; Degenerative cervical radiculopathy; ASD; Adjacent Segment Disease; Adjacent Level Disease
MeSH Terms: conditions — Radiculopathy; Spinal Cord Compression; Spinal Cord Diseases; Spondylosis; Klippel-Feil Syndrome | interventions — Gene Fusion; Arthroplasty

STUDY DESIGN:
Intervention Model Description: Prospective Single-blind Randomised Controlled Trial with computer randomization in a 1:1 ratio
Who Masked: Participant
Masking Description: Participants will be blinded until one-year after allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACDF (Active Comparator): Anterior cervical discectomy and fusion.
  Interventions: Procedure: ACDF
- ACDA (Experimental): Anterior cervical discectomy with arthroplasty.
  Interventions: Procedure: ACDA

INTERVENTIONS:
Procedure: ACDF — Standard operative treatment for anterior cervical discectomy. Through a right or left-sided approach the disc space contents are resected. The endplates are prepared with curettes and the disc space contents are removed. The posterior longitudinal ligament is opened. The dura is visualized to ensure adequate decompression. A cage is implanted in the disc space. The disc removal and cage implantation can be performed at a single level or at multiple levels. The wound is closed in layers, after a prevertebral wound drain is placed.
  Other Names: Anterior Cervical Discectomy and Fusion
  Arms: ACDF
Procedure: ACDA — The start of the procedure is the same as in the ACDF group. After the discectomy, a cervical disc prosthesis is placed in the disc space instead of a cage, in accordance with the manufacturer's protocol for implantation and endplate preparation. The disc removal and arthrodesis implantation can be performed at a single level or at multiple levels. Wound closure is similar to the ACDF procedure.
  Other Names: Anterior Cervical Discectomy and arthroplasty
  Arms: ACDA

SUMMARY:
To date, no consensus exists on which anterior surgical technique is more cost-effective to treat cervical degenerative disc disease (CDDD). The most commonly used surgical treatment for patients with single- or multilevel symptomatic CDDD is anterior cervical discectomy with fusion (ACDF). However, new complaints of radiculopathy and/or myelopathy commonly develop at adjacent levels, also known as clinical adjacent segment pathology (CASP). It remains unknown to what extent kinematics, surgery-induced fusion and natural history of disease play a role in its development. Anterior cervical discectomy with arthroplasty (ACDA) is thought to reduce the incidence of CASP by preserving motion in the operated segment. ACDA is often discouraged as the implant costs are higher whilst the clinical outcomes are similar to ACDF. However, preventing CASP might be a reason for ACDA to be a more cost-effective technique in the long-term.

In this randomized controlled trial patients will be randomized to receive ACDF or ACDA in a 1:1 ratio. Adult patients with single- or multi-level CDDD and symptoms of radiculopathy and/or myelopathy will be included. The primary outcome is cost-effectiveness and cost-utility of both techniques from a societal perspective. Secondary objectives are the differences in clinical and radiological outcomes between the two techniques, as well as the qualitative process surrounding anterior decompression surgery. All outcomes will be measured at baseline and every 6 months till 4 years postoperatively.

High quality evidence regarding the cost-effectiveness of both ACDA and ACDF is lacking, to date no prospective trials from a societal perspective exist. Considering the ageing of the population and the rising healthcare costs, the need for a solid clinical cost-effectiveness trial addressing this question is high.

DETAILED DESCRIPTION:
Cervical degenerative disc disease (CDDD) is the degeneration of a cervical intervertebral disc and/or the adjoining vertebral bodies, resulting in clinical symptoms of cervical radiculopathy, myelopathy, myeloradiculopathy, and axial pain. The incidence of degenerative pathologies is significantly increasing as the population of elderly is rising. Currently, generalized spinal disc degeneration occurs in more than 90% of adults past the 5th decade of life.This age group now represents 32.8% of the population in Europe and is projected to reach 40.6% by 2050. In the next 20 years a significant increase in anterior cervical decompression surgeries is predicted in those aged 45-54, mainly affecting the working population. Complaints of radiculopathy and/or myelopathy lead to restrictions in daily life and loss of professional capability, resulting in absenteeism. Societal healthcare costs are therefore significantly affected by CDDD. The healthcare costs are driven up further when patients require surgical treatment, in combination with associated hospitalization and rehabilitation. To date, no consensus exists on which anterior surgical technique is more cost-effective to treat CDDD with radiculopathy and/or myelopathy.

One of the most common procedures for treating patients with single- or multilevel CDDD is anterior cervical discectomy with fusion (ACDF). ACDF results in fusion in 95-100%. The primary goal of ACD(F) is the relief of symptoms of radiculopathy and/or myelopathy through decompression of neural structures. Fusion in itself is not a requisite to reach this goal. In our center, ACDF with stand-alone cages is the standard procedure for CDDD. Plate-constructs are only used on indication. A common concern regarding ACDF with stand-alone cages is the occurrence of cage subsidence. In our retrospective cohort of 673 patients, only 1 patient required additional surgery due to subsidence (0.15%) [unpublished data]. Axial pain alone is not considered an indication for surgical treatment. Good short-term clinical results are achieved for both radiculopathy and myelopathy. Clinical results are independent from the technique used, and independent from occurrence of fusion. However, patient-reported satisfaction gradually decreases in the years following surgery. This is thought to be the consequence of the development of new complaints due to degenerative changes at a segment adjacent to the site of the index surgery, also known as adjacent segment pathology (ASP).

A recent consensus proposes a distinct definition of radiologic adjacent segment pathology (RASP) and clinical adjacent segment pathology (CASP). CASP occurs at an estimated cumulative rate of 1.6% to 4.2% per year after ACDF, however, a wide variety in incidence is reported in literature. About 50-75% of the patients that develop CASP require additional adjacent segment surgery. In our retrospective cohort, we observed a rate of 2.1% CASP per year, with an additional adjacent segment surgery rate of 1.5% per year. Moreover, we found that half of these patients undergo additional surgery for CASP within 2.5 years, which suggests a peak incidence in the first years following index surgery. The underlying mechanism of ASP remains a matter of debate. Besides natural degeneration, compensation for the loss of motion in the fused segment is thought to cause overstraining of the adjacent segments. Altered cervical sagittal alignment is also thought to be of importance in the accelerated development of CASP. Higher rates of CASP are observed after ACD, concomitant with an increased segmental kyphosis at the index level. Unlike ACD, ACDF with plate-constructs restore cervical sagittal lordosis. However, a higher rate of ASP is observed in those with plate-constructs in comparison to ACDF with stand-alone cages. The higher rate of ASP after ACDF with plate-constructs might be explained by strain on the adjacent segments by the plate, or more extensive surgical preparation for installing the plate increasing the chance on destruction of the adjacent level. Another contributing factor might be the occurrence of subsidence of the plate-construct into the adjacent segment. Disc height at the adjacent segments is found to be significantly decreased in those with plate-constructs, which supports this theory. It remains unknown to what extent altered cervical motion influences the development of ASP.

Anterior cervical discectomy with arthroplasty (ACDA) was developed to reduce the incidence of CASP by preserving motion in the operated segment. Previously conducted research in patients with radiculopathy and/or myelopathy has shown no significant differences in clinical or radiological outcomes amongst ACDA and ACD(F). A meta-analysis found better neurological outcomes in patients with myelopathy after ACDA, in contrast to the pre-existing notion that ACDA leads to less favorable outcomes in myelopathy due to micro-trauma caused by preserved mobility. Moreover, additional adjacent segment surgery rates are significantly lower for ACDA, both for single- and multilevel surgeries. The difference in additional adjacent segment surgery rates between ACDA and ACDF expands exponentially with a longer-follow-up time. ACDA is often discouraged as the implant costs are higher than those for ACDF whilst clinical outcomes are similar. However, preventing new complaints and additional surgeries due to CASP might be a reason for ACDA to be a more cost-effective technique in the long-term. A systematic review of economic evaluations in anterior cervical decompression surgery was conducted by our research group. The majority of studies report ACDA to be the most cost-effective technique despite higher implant costs. Literature was however strongly heterogeneous and of low quality.

In conclusion, there is increasing evidence suggesting that ACDA might be the more cost-effective technique because of a reduced risk on CASP and associated additional surgery rates, compared to ACD(F). High quality evidence regarding the cost-effectiveness of both ACDA and ACDF is lacking, especially in Europe. Therefore, the need for a solid clinical cost-effectiveness trial addressing this question is high.

ELIGIBILITY:
Inclusion Criteria:

* Indication for anterior cervical decompression surgery.
* Single- or multilevel CDDD between C3 and C7.
* Symptoms of myelopathy, radiculopathy, or myeloradiculopathy.
* In case of pure radiculopathy: refractory to at least 6 weeks of conservative therapy.
* In case of myelopathy: symptomatic myelopathy.
* Patients ≥ 18 years of age.

Exclusion criteria

* Indication for (additional) posterior surgical approach.
* Indication for additional stabilization of the pathological segment by a plate.
* Previous ventral surgery of the cervical spine.
* Traumatic origin of the compression.
* Previous radiotherapy of the cervical spine.
* Metabolic bone disease.
* Inflammatory spinal disease: e.g., Bechterew's disease, Forestier's disease.
* Infection of the cervical spine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Costs | 4 years
  Costs will be determined from a societal perspective.
  Validated cost questionnaires for societal costs, including medical consumption, both paid and unpaid loss of productivity for patients. :
  * Productivity Cost Questionnaire (iPCQ) for measuring productivity loss for work loss (paid and unpaid). Consists of 7 questions.
  * the Medical Consumption Questionnaire (iMCQ) for measuring medical consumption, especially designed for the Dutch health care environment. Consists of 14 questions.
  Informal caregivers will be asked to fill out the Limited Valuation of Informal Care Questionnaire (iVICQ):
  * informal care giver (ICG) productivity loss for work loss (paid and unpaid)
  * Care-related Quality of Life instrument (CarerQol-7D).
  * The Self-Rated Burden scale (SRB), a horizontal 'visual-analog scale' to determine the subjective burden of the caregiver on a scale from 0 (not heavy) to 10 (very heavy).
Effectiveness | 4 years
  In the CUA, the Incremental Cost-Effectiveness Ratio (ICER) will be expressed as the incremental costs per QALY.
  Quality Adjusted Life Years (QALYs) will be determined by Generic Quality of Life assessed based on the EuroQol utility scores (EQ-5D-5L). The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

SECONDARY OUTCOMES:
CASP | 4 years
  The rate of clinical adjacent segment pathology and associated additional surgeries will be assessed.
Radiological Outcomes | 1 year
  At 3 time points; pre-operatively, directly post-operative and one-year post-operative.
  * Pre-operative imaging will assess baseline degeneration according to the Kellgren-Lawrence Score, cervical sagittal alignment and baseline disc height. Moreover, a full sagittal spine X-ray will be made to assess pre-operative global balance according to the odontoid-hip axis.
  * Post-operative: A standard cervical spine X-ray to assess the position of the implant, subsidence and cervical sagittal alignment.
  * 1 year post-operative cervical spine X-rays will be made. A standard cervical spine X-ray will be made to assess fusion, cage subsidence, adjacent segment degeneration (KS), adjacent segment disc height and alignment. A flexion and extension X-ray will be made to assess movement.
Neck Disability Index (NDI). | 4 years
  It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each question is scored on a 0-5 scale, where 0 is no disability and 5 is the maximal disability possible
Visual Analogue Scale (VAS) for neck and arm pain. | 4 years
  Visual Analogue Scale (VAS) for neck and arm pain. Neck and arm pain are assessed separately on a horizontal 10 cm visual scale, varying from 0 cm (no pain) to 10 cm (worst pain imaginable)
Hospital Anxiety Depression Scale (HADS) | 4 years
  A fourteen-item scale, to determine the anxiety and depression level. Consisting of a 7-item depression scale and a 7-item anxiety scale. The score ranges from 0-21 with a high score being indicative for depression/anxiety (≥ 8)
modified Japanese Orthopedic Association score (mJOA) | 4 years
  modified Japanese Orthopedic Association score (mJOA) for myelopathy. patients. An investigator-administered tool used to evaluate neurological function in patients with cervical myelopathy. It is an 18-point scale that addresses upper (5 points) and lower extremity (7 points) motor function, sensation (3 points) and micturition (3 points). A score of 18 reflects no neurological deficits whereas a lower score indicates a greater degree of disability and functional impairment
Process Evaluation | 4 years
  Moreover, a process evaluation will be performed to determine the underlying values, needs, impacts and preferences of people with CDDD. The focus will be experiences and opinions of patients, caregivers, and professionals concerning the process surrounding ACDA and ACDF. A process evaluation might also identify gaps or limitations in published research with regards to important outcomes to those with lived experience. A qualitative analysis will be performed according to the framework provided by Saunders et al.

CONTACTS AND LOCATIONS:
Overall Officials: Anouk Smeets, MD, PhD, Professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Zuyderland Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Radhakrishnan K, Litchy WJ, O'Fallon WM, Kurland LT. Epidemiology of cervical radiculopathy. A population-based study from Rochester, Minnesota, 1976 through 1990. Brain. 1994 Apr;117 ( Pt 2):325-35. doi: 10.1093/brain/117.2.325. PMID 8186959
- [Background] Salemi G, Savettieri G, Meneghini F, Di Benedetto ME, Ragonese P, Morgante L, Reggio A, Patti F, Grigoletto F, Di Perri R. Prevalence of cervical spondylotic radiculopathy: a door-to-door survey in a Sicilian municipality. Acta Neurol Scand. 1996 Feb-Mar;93(2-3):184-8. doi: 10.1111/j.1600-0404.1996.tb00196.x. PMID 8741140
- [Background] McCartney S, Baskerville R, Blagg S, McCartney D. Cervical radiculopathy and cervical myelopathy: diagnosis and management in primary care. Br J Gen Pract. 2018 Jan;68(666):44-46. doi: 10.3399/bjgp17X694361. No abstract available. PMID 29284641
- [Background] Boogaarts HD, Bartels RH. Prevalence of cervical spondylotic myelopathy. Eur Spine J. 2015 Apr;24 Suppl 2:139-41. doi: 10.1007/s00586-013-2781-x. Epub 2013 Apr 25. PMID 23616201
- [Background] Kuijper B, Tans JT, Schimsheimer RJ, van der Kallen BF, Beelen A, Nollet F, de Visser M. Degenerative cervical radiculopathy: diagnosis and conservative treatment. A review. Eur J Neurol. 2009 Jan;16(1):15-20. doi: 10.1111/j.1468-1331.2008.02365.x. PMID 19087147
- [Background] Saal JS, Saal JA, Yurth EF. Nonoperative management of herniated cervical intervertebral disc with radiculopathy. Spine (Phila Pa 1976). 1996 Aug 15;21(16):1877-83. doi: 10.1097/00007632-199608150-00008. PMID 8875719
- [Background] Fehlings MG, Tetreault LA, Riew KD, Middleton JW, Aarabi B, Arnold PM, Brodke DS, Burns AS, Carette S, Chen R, Chiba K, Dettori JR, Furlan JC, Harrop JS, Holly LT, Kalsi-Ryan S, Kotter M, Kwon BK, Martin AR, Milligan J, Nakashima H, Nagoshi N, Rhee J, Singh A, Skelly AC, Sodhi S, Wilson JR, Yee A, Wang JC. A Clinical Practice Guideline for the Management of Patients With Degenerative Cervical Myelopathy: Recommendations for Patients With Mild, Moderate, and Severe Disease and Nonmyelopathic Patients With Evidence of Cord Compression. Global Spine J. 2017 Sep;7(3 Suppl):70S-83S. doi: 10.1177/2192568217701914. Epub 2017 Sep 5. PMID 29164035
- [Background] Badhiwala JH, Wilson JR. The Natural History of Degenerative Cervical Myelopathy. Neurosurg Clin N Am. 2018 Jan;29(1):21-32. doi: 10.1016/j.nec.2017.09.002. Epub 2017 Oct 27. PMID 29173433
- [Background] Dowd GC, Wirth FP. Anterior cervical discectomy: is fusion necessary? J Neurosurg. 1999 Jan;90(1 Suppl):8-12. doi: 10.3171/spi.1999.90.1.0008. PMID 10413119
- [Background] Donk RD, Verbeek ALM, Verhagen WIM, Groenewoud H, Hosman AJF, Bartels RHMA. What's the best surgical treatment for patients with cervical radiculopathy due to single-level degenerative disease? A randomized controlled trial. PLoS One. 2017 Aug 29;12(8):e0183603. doi: 10.1371/journal.pone.0183603. eCollection 2017. PMID 28850600
- [Background] Nandoe Tewarie RD, Bartels RH, Peul WC. Long-term outcome after anterior cervical discectomy without fusion. Eur Spine J. 2007 Sep;16(9):1411-6. doi: 10.1007/s00586-007-0309-y. Epub 2007 Jan 30. PMID 17262184
- [Background] Hilibrand AS, Carlson GD, Palumbo MA, Jones PK, Bohlman HH. Radiculopathy and myelopathy at segments adjacent to the site of a previous anterior cervical arthrodesis. J Bone Joint Surg Am. 1999 Apr;81(4):519-28. doi: 10.2106/00004623-199904000-00009. PMID 10225797
- [Background] Eck JC, Humphreys SC, Lim TH, Jeong ST, Kim JG, Hodges SD, An HS. Biomechanical study on the effect of cervical spine fusion on adjacent-level intradiscal pressure and segmental motion. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2431-4. doi: 10.1097/00007632-200211150-00003. PMID 12435970
- [Background] Boselie TF, Willems PC, van Mameren H, de Bie RA, Benzel EC, van Santbrink H. Arthroplasty versus fusion in single-level cervical degenerative disc disease: a Cochrane review. Spine (Phila Pa 1976). 2013 Aug 1;38(17):E1096-107. doi: 10.1097/BRS.0b013e3182994a32. PMID 23656959
- [Background] Boselie TF, van Santbrink H. Arthroplasty in cervical degenerative disc disease: fulfilling its long-term promise? J Spine Surg. 2016 Dec;2(4):359-361. doi: 10.21037/jss.2016.12.01. No abstract available. PMID 28097260
- [Background] Joaquim AF, Riew KD. Multilevel cervical arthroplasty: current evidence. A systematic review. Neurosurg Focus. 2017 Feb;42(2):E4. doi: 10.3171/2016.10.FOCUS16354. PMID 28142256
- [Background] Radcliff K, Davis RJ, Hisey MS, Nunley PD, Hoffman GA, Jackson RJ, Bae HW, Albert T, Coric D. Long-term Evaluation of Cervical Disc Arthroplasty with the Mobi-C(c) Cervical Disc: A Randomized, Prospective, Multicenter Clinical Trial with Seven-Year Follow-up. Int J Spine Surg. 2017 Nov 28;11(4):31. doi: 10.14444/4031. eCollection 2017. PMID 29372135
- [Background] Davis RJ, Kim KD, Hisey MS, Hoffman GA, Bae HW, Gaede SE, Rashbaum RF, Nunley PD, Peterson DL, Stokes JK. Cervical total disc replacement with the Mobi-C cervical artificial disc compared with anterior discectomy and fusion for treatment of 2-level symptomatic degenerative disc disease: a prospective, randomized, controlled multicenter clinical trial: clinical article. J Neurosurg Spine. 2013 Nov;19(5):532-45. doi: 10.3171/2013.6.SPINE12527. Epub 2013 Sep 6. PMID 24010901
- [Background] Arts MP, Brand R, van den Akker E, Koes BW, Peul WC. The NEtherlands Cervical Kinematics (NECK) trial. Cost-effectiveness of anterior cervical discectomy with or without interbody fusion and arthroplasty in the treatment of cervical disc herniation; a double-blind randomised multicenter study. BMC Musculoskelet Disord. 2010 Jun 16;11:122. doi: 10.1186/1471-2474-11-122. PMID 20553591
- [Background] Bartels RH, Donk R, van der Wilt GJ, Grotenhuis JA, Venderink D. Design of the PROCON trial: a prospective, randomized multi-center study comparing cervical anterior discectomy without fusion, with fusion or with arthroplasty. BMC Musculoskelet Disord. 2006 Nov 10;7:85. doi: 10.1186/1471-2474-7-85. PMID 17096851
- [Background] Bartels RH, Donk R, Verbeek AL. No justification for cervical disk prostheses in clinical practice: a meta-analysis of randomized controlled trials. Neurosurgery. 2010 Jun;66(6):1153-60; discussion 1160. doi: 10.1227/01.NEU.0000369189.09182.5F. PMID 20421840
- [Background] Radcliff K, Zigler J, Zigler J. Costs of cervical disc replacement versus anterior cervical discectomy and fusion for treatment of single-level cervical disc disease: an analysis of the Blue Health Intelligence database for acute and long-term costs and complications. Spine (Phila Pa 1976). 2015 Apr 15;40(8):521-9. doi: 10.1097/BRS.0000000000000822. PMID 25868092
- [Background] M Versteegh M, M Vermeulen K, M A A Evers S, de Wit GA, Prenger R, A Stolk E. Dutch Tariff for the Five-Level Version of EQ-5D. Value Health. 2016 Jun;19(4):343-52. doi: 10.1016/j.jval.2016.01.003. Epub 2016 Mar 30. PMID 27325326
- [Background] Nederland Z. Guideline for economic evaluations in healthcare. 2016.
- [Background] Bouwmans C, Krol M, Severens H, Koopmanschap M, Brouwer W, Hakkaart-van Roijen L. The iMTA Productivity Cost Questionnaire: A Standardized Instrument for Measuring and Valuing Health-Related Productivity Losses. Value Health. 2015 Sep;18(6):753-8. doi: 10.1016/j.jval.2015.05.009. Epub 2015 Aug 20. PMID 26409601
- [Background] C. Bouwmans et al. . Rotterdam: iMTA EUR, 2013. Handleiding iMTA Medical Cost Questionnaire (iMCQ). Value Heal. 2013;18:753-758.
- [Background] Hoefman RJ VEN, Brouwer WBF. iMTA Valuation of Informal Care Questionnaire (iVICQ). Version 1.0. 2011
- [Background] Vernon H. The Neck Disability Index: state-of-the-art, 1991-2008. J Manipulative Physiol Ther. 2008 Sep;31(7):491-502. doi: 10.1016/j.jmpt.2008.08.006. PMID 18803999
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Spinhoven P, Ormel J, Sloekers PP, Kempen GI, Speckens AE, Van Hemert AM. A validation study of the Hospital Anxiety and Depression Scale (HADS) in different groups of Dutch subjects. Psychol Med. 1997 Mar;27(2):363-70. doi: 10.1017/s0033291796004382. PMID 9089829
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Tetreault L, Kopjar B, Nouri A, Arnold P, Barbagallo G, Bartels R, Qiang Z, Singh A, Zileli M, Vaccaro A, Fehlings MG. The modified Japanese Orthopaedic Association scale: establishing criteria for mild, moderate and severe impairment in patients with degenerative cervical myelopathy. Eur Spine J. 2017 Jan;26(1):78-84. doi: 10.1007/s00586-016-4660-8. Epub 2016 Jun 24. PMID 27342612
- [Background] Saunders RP, Evans MH, Joshi P. Developing a process-evaluation plan for assessing health promotion program implementation: a how-to guide. Health Promot Pract. 2005 Apr;6(2):134-47. doi: 10.1177/1524839904273387. PMID 15855283
- [Background] Cepoiu-Martin M, Faris P, Lorenzetti D, Prefontaine E, Noseworthy T, Sutherland L. Artificial cervical disc arthroplasty: a systematic review. Spine (Phila Pa 1976). 2011 Dec 1;36(25):E1623-33. doi: 10.1097/BRS.0b013e3182163814. PMID 22101705
- [Background] McAfee PC, Reah C, Gilder K, Eisermann L, Cunningham B. A meta-analysis of comparative outcomes following cervical arthroplasty or anterior cervical fusion: results from 4 prospective multicenter randomized clinical trials and up to 1226 patients. Spine (Phila Pa 1976). 2012 May 15;37(11):943-52. doi: 10.1097/BRS.0b013e31823da169. PMID 22037535
- [Background] Upadhyaya CD, Wu JC, Trost G, Haid RW, Traynelis VC, Tay B, Coric D, Mummaneni PV. Analysis of the three United States Food and Drug Administration investigational device exemption cervical arthroplasty trials. J Neurosurg Spine. 2012 Mar;16(3):216-28. doi: 10.3171/2011.6.SPINE10623. Epub 2011 Dec 23. PMID 22195608
- [Background] Jiang H, Zhu Z, Qiu Y, Qian B, Qiu X, Ji M. Cervical disc arthroplasty versus fusion for single-level symptomatic cervical disc disease: a meta-analysis of randomized controlled trials. Arch Orthop Trauma Surg. 2012 Feb;132(2):141-51. doi: 10.1007/s00402-011-1401-7. Epub 2011 Oct 9. PMID 21984009
- [Background] Yu L, Song Y, Yang X, Lv C. Systematic review and meta-analysis of randomized controlled trials: comparison of total disk replacement with anterior cervical decompression and fusion. Orthopedics. 2011 Oct 5;34(10):e651-8. doi: 10.3928/01477447-20110826-09. PMID 21956061
- [Background] Hilibrand AS, Robbins M. Adjacent segment degeneration and adjacent segment disease: the consequences of spinal fusion? Spine J. 2004 Nov-Dec;4(6 Suppl):190S-194S. doi: 10.1016/j.spinee.2004.07.007. PMID 15541666
- [Background] Powell JW, Sasso RC, Metcalf NH, Anderson PA, Hipp JA. Quality of spinal motion with cervical disk arthroplasty: computer-aided radiographic analysis. J Spinal Disord Tech. 2010 Apr;23(2):89-95. doi: 10.1097/BSD.0b013e3181991413. PMID 20051921
- [Background] Sasso RC, Best NM. Cervical kinematics after fusion and bryan disc arthroplasty. J Spinal Disord Tech. 2008 Feb;21(1):19-22. doi: 10.1097/BSD.0b013e3180500778. PMID 18418131
- [Background] Sasso RC, Best NM, Metcalf NH, Anderson PA. Motion analysis of bryan cervical disc arthroplasty versus anterior discectomy and fusion: results from a prospective, randomized, multicenter, clinical trial. J Spinal Disord Tech. 2008 Aug;21(6):393-9. doi: 10.1097/BSD.0b013e318150d121. PMID 18679092
- [Background] Nabhan A, Steudel WI, Nabhan A, Pape D, Ishak B. Segmental kinematics and adjacent level degeneration following disc replacement versus fusion: RCT with three years of follow-up. J Long Term Eff Med Implants. 2007;17(3):229-36. doi: 10.1615/jlongtermeffmedimplants.v17.i3.60. PMID 19023947
- [Background] Park DK, Lin EL, Phillips FM. Index and adjacent level kinematics after cervical disc replacement and anterior fusion: in vivo quantitative radiographic analysis. Spine (Phila Pa 1976). 2011 Apr 20;36(9):721-30. doi: 10.1097/BRS.0b013e3181df10fc. PMID 20543765
- [Background] Boselie TF, Willems PC, van Mameren H, de Bie R, Benzel EC, van Santbrink H. Arthroplasty versus fusion in single-level cervical degenerative disc disease. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD009173. doi: 10.1002/14651858.CD009173.pub2. PMID 22972137
- [Background] Punt I, Baxter R, van Ooij A, Willems P, van Rhijn L, Kurtz S, Steinbeck M. Submicron sized ultra-high molecular weight polyethylene wear particle analysis from revised SB Charite III total disc replacements. Acta Biomater. 2011 Sep;7(9):3404-11. doi: 10.1016/j.actbio.2011.05.010. Epub 2011 May 20. PMID 21621656
- [Background] Punt IM, Austen S, Cleutjens JP, Kurtz SM, ten Broeke RH, van Rhijn LW, Willems PC, van Ooij A. Are periprosthetic tissue reactions observed after revision of total disc replacement comparable to the reactions observed after total hip or knee revision surgery? Spine (Phila Pa 1976). 2012 Jan 15;37(2):150-9. doi: 10.1097/BRS.0b013e3182154c22. PMID 21336235
- [Derived] Schuermans VNE, Smeets AYJM, Boselie TFM, Candel MJJM, Curfs I, Evers SMAA, Van Santbrink H. Research protocol: Cervical Arthroplasty Cost Effectiveness Study (CACES): economic evaluation of anterior cervical discectomy with arthroplasty (ACDA) versus anterior cervical discectomy with fusion (ACDF) in the surgical treatment of cervical degenerative disc disease - a randomized controlled trial. Trials. 2022 Aug 26;23(1):715. doi: 10.1186/s13063-022-06574-5. PMID 36028916